CLINICAL TRIAL: NCT02524795
Title: Omega 3 Fatty Acids, Inflammatory Status and Biochemical Markers of Patients With Systemic Lupus Erythematosus: a Pilot Study
Brief Title: Omega 3 Fatty Acids and Systemic Lupus Erythematosus
Acronym: OM3LES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Cristina Costa Duarte Lanna, MD, PhD, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LES-001-O3
Record Dates: First submitted 2015-07-08; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Omega 3, Cytokines, Adipokines, Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hiomega-3 supplement (Experimental): Patients in the study group received, throughout 12 weeks, two tablets per day of omega-3 fatty acids (540mg of EPA and DHA of 100mg; Hiomega-3 supplement of Naturalis® company). Participants were seen at baseline (T0) and at week 12 (T1) for clinical, laboratory and nutritional assessment.
  Variables measured at each visit included: disease activity index, using the Systemic Lupus Disease Activity Index (SLEDAI-2k)16; damage index (Systemic Lupus International Collaboration Clinics/American College of Rheumatology damage index - SLICC/ACR)17; fasting lipid and glucose proﬁle; standard laboratory tests to assess SLE ; cytokines (IL-6, IL-10), adipokines (leptin, adiponectin) C-reactive protein (CRP), nutritional assessment, and in use medications.
  Interventions: Dietary Supplement: Hiomega-3 supplement of Naturalis® company -
- Control group (No Intervention): Patients in the control group did not receive the nutrient nor any kind of placebo. They were seen at baseline (T0) and at week 12 (T1) for clinical, laboratory and nutritional assessment.
  Variables measured at each visit included: disease activity index, using the Systemic Lupus Disease Activity Index (SLEDAI-2k)16; damage index (Systemic Lupus International Collaboration Clinics/American College of Rheumatology damage index - SLICC/ACR)17; fasting lipid and glucose proﬁle; standard laboratory tests to assess SLE ; cytokines (IL-6, IL-10), adipokines (leptin, adiponectin) C-reactive protein (CRP), nutritional assessment, and in use medications.

INTERVENTIONS:
Dietary Supplement: Hiomega-3 supplement of Naturalis® company - — Patients (N=22) were seen at baseline (T0) and at week 12 (T1) for clinical, laboratory and nutritional assessment, and were contacted by telephone in week 6 to check on compliance and any adverse events. Patients received, throughout 12 weeks, two tablets per day of omega-3 fatty acids (540mg of EPA and DHA of 100mg; Hiomega-3 supplement of Naturalis® company - registered in the National Health Department number 4.1480.0006.001-4). All participants were instructed not to take omega-3 rich foods during the study period.
  Arms: Hiomega-3 supplement

SUMMARY:
Omega-3 fatty acids have been considered anti-inflammatory lipids based on data from epidemiological studies of Greenland Eskimos whose diet is rich in fish, sources of polyunsaturated fatty acids.

Fatty acids from the omega-3 family [mainly the α-linolenic acid, eicosapentaenoic (EPA) and docosahexaenoic (DHA)], as well as those of the omega-6 family [represented mainly by linoleic acid and arachidonic acid (AA)] are essential for the synthesis of eicosanoids, prostaglandins, leukotrienes, thromboxanes and other oxidative factors, major mediators and regulators of inflammation.

Systemic lupus erythematosus (SLE) is an inflammatory autoimmune disease characterized by the loss of balance of cellular immunoregulation and increased levels of circulating inflammatory mediators.Thus, omega-3 supplementation could represent additional therapy for individuals with SLE.

The aim of this study was to investigate the effects of omega-3 fatty acids on circulating levels of inflammatory and biochemical markers in women with SLE.

DETAILED DESCRIPTION:
This is a pilot clinical trial of omega-3-polyunsaturated fatty acids carried out in SLE patients followed at the Rheumatology Unit of Hospital das Clínicas, Universidade Federal de Minas Gerais, UFMG.

Female patients who met the revised American College of Rheumatology (ACR) classiﬁcation criteria for SLE (1982/1997)15, age over 18 years old and below 60 years old, who were taking stable doses of medications for the SLE treatment in the last three months were included. Exclusion criteria were the following: pregnancy, disease duration of less than one year, allergy to ﬁsh, ﬁsh oil or any omega-3 product, omega-3 use within the previous six months and diagnosis of diabetes mellitus, liver disease, chronic renal failure, any type of infection at enrollment and/or throughout the study.

A 12 week pilot clinical trial of omega-3 fatty acid supplementation was conducted. Participants were seen at baseline (T0) and at week 12 (T1) for clinical, laboratory and nutritional assessment. Participants were also contacted by telephone in week 6 to check on compliance and any adverse events. The patients were randomized into one of two groups in a 1:1 ratio. Patients in the study group received, throughout 12 weeks, two tablets per day of omega-3 fatty acids (540mg of EPA and DHA of 100mg; Hiomega-3 supplement of Naturalis® company - registered in the National Health Department number 4.1480.0006.001-4). Patients in the control group did not receive the nutrient nor any kind of placebo. All participants were instructed not to take omega-3 rich foods during the study period. The researcher (FMMS) who did clinical assessment and the inflammatory and biochemical data assessment was blind to randomization and intervention.

Variables measured at each visit included: disease activity index, using the Systemic Lupus Disease Activity Index (SLEDAI-2k)16; damage index (Systemic Lupus International Collaboration Clinics/American College of Rheumatology damage index - SLICC/ACR)17; fasting lipid and glucose proﬁle; standard laboratory tests to assess SLE (red and white blood count, platelet count, creatinine, urinalysis, urine protein/creatinine ratio, anti-dsDNA, anticardiolipin, C3 and C4 levels); cytokines (IL-6, IL-10), adipokines (leptin, adiponectin) C-reactive protein (CRP), nutritional assessment, and in use medications.

ELIGIBILITY:
Inclusion Criteria: 1-Diagnosis of lupus according to American College of Rheumatology (ACR) classiﬁcation criteria for SLE (1982/1997)

* Taking stable doses of medications for the SLE treatment in the last three months.

Exclusion Criteria:

* pregnancy, disease duration of less than one year, allergy to ﬁsh, ﬁsh oil or any omega-3 product, omega-3 use within the previous six months and diagnosis of diabetes mellitus, liver disease, chronic renal failure, any type of infection at enrollment and/or throughout the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Variations of serum cytokines related to omega 3 treatment | Cytokines measurement on T0 (baseline) and T1 (after 12 weeks)
  The primary outcomes was median (interquartile range, IQR) variations [ΔV=pre-Treatment (T0) minus post-treatment (T1) concentrations] of serum cytokines (IL6 e IL 10) after 12 weeks of treatment between groups.
Variations of serum adipokines related to omega 3 treatment | Adipokines measurement on T0 (baseline) and T1 (after 12 weeks)
  The primary outcomes was median (interquartile range, IQR) variations [ΔV=pre-Treatment (T0) minus post-treatment (T1) concentrations] of serum adipokines (leptin and adiponectin) after 12 weeks of treatment between groups.
Variations of serum C reactive protein related to omega 3 treatment | C reactive protein measurement on T0 (baseline) and T1 (after 12 weeks)
  The primary outcomes was median (interquartile range, IQR) variations [ΔV=pre-Treatment (T0) minus post-treatment (T1) concentrations] of serum C reactive protein after 12 weeks of treatment between groups.

SECONDARY OUTCOMES:
Variations of biochemical markers related to omega 3 treatment | Biochemical markers measurement on T0 (baseline) and T1 (after 12 weeks)
  The primary outcomes was median (interquartile range, IQR) variations [ΔV=pre-Treatment (T0) minus post-treatment (T1) concentrations] of biochemical markers (glucose and lipidis) after 12 weeks of treatment between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Isabel TD Correia, PhD, Principal Investigator — Federal University of Minas Gerais

REFERENCES:
- [Derived] Curado Borges M, de Miranda Moura Dos Santos F, Weiss Telles R, Melo de Andrade MV, Toulson Davisson Correia MI, Lanna CCD. Omega-3 fatty acids, inflammatory status and biochemical markers of patients with systemic lupus erythematosus: a pilot study. Rev Bras Reumatol Engl Ed. 2017 Nov-Dec;57(6):526-534. doi: 10.1016/j.rbre.2016.09.014. Epub 2016 Oct 22. English, Portuguese. PMID 29173690